CLINICAL TRIAL: NCT02963025
Title: PROtective Ventilation With High Versus Low PEEP During One-lung Ventilation for THORacic Surgery PROTHOR: A Randomized Controlled Trial
Brief Title: Protective Ventilation With High Versus Low PEEP During One-lung Ventilation for Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Istanbul University (Other); European Society of Anaesthesiology and Intensive Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK 392092016
Record Dates: First submitted 2016-11-10; First posted 2016-11-15 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: One-Lung Ventilation
Keywords: Mechanical ventilation; positive end-expiratory pressure; recruitment maneuver; one-lung ventilation; thoracic surgery; postoperative pulmonary complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- THE HIGHER PEEP LEVEL (Other): Mechanical ventilation with VT of 5 ml/kg PBW and the level of PEEP at 10 cmH2O with lung recruitment maneuvers
  Interventions: Procedure: PEEP level; Procedure: Use of recruitment maneuvers
- THE LOWER PEEP LEVEL (Other): Mechanical ventilation with VT of 5 ml/kg PBW and the level of PEEP at 5 cmH2O without lung recruitment maneuvers
  Interventions: Procedure: PEEP level

INTERVENTIONS:
Procedure: PEEP level
Procedure: Use of recruitment maneuvers
  Arms: THE HIGHER PEEP LEVEL

SUMMARY:
One-lung ventilation (OLV) with resting of the contralateral lung may be required to allow or facilitate thoracic surgery. However, OLV can result in severe hypoxemia, requiring a mechanical ventilation approach that is able to maintain adequate gas exchange, while protecting the lungs against postoperative pulmonary complications (PPCs). During OLV, the use of lower tidal volumes is helpful to avoid over-distension, but can result in increased atelectasis and repetitive collapse-and-reopening of lung units, particularly at low levels of positive end-expiratory pressure (PEEP).

Anesthesiologists inconsistently use PEEP and recruitment maneuvers (RM) in the hope that this may improve oxygenation and protect against PPC. Up to now, it is not known whether high levels of PEEP combined with RM are superior to lower PEEP without RM for protection against PPCs during OLV.

Hypothesis: An intra-operative ventilation strategy using higher levels of PEEP and recruitment maneuvers, as compared to ventilation with lower levels of PEEP without recruitment maneuvers, prevents postoperative pulmonary complications in patients undergoing thoracic surgery under standardized one-lung ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open thoracic or video-assisted thoracoscopic surgery under general anesthesia requiring OLV (no emergency surgery)
* BMI < 35 kg/m2
* age ≥ 18 years
* expected duration of surgery > 60 min
* planned lung separation with double lumen tube (DLT, not for study purpose only)
* most of ventilation time during surgery expected to be in OLV

Exclusion Criteria:

* COPD GOLD grades III and IV, lung fibrosis, documented bullae, severe emphysema, pneumothorax
* uncontrolled asthma
* Heart failure NYHA Grade 3 and 4, Coronary Heart Disease CCS Grade 3 and 4
* previous lung surgery
* documented pulmonary arterial hypertension >25mmHg MPAP at rest or > 40 mmHg syst. (estimated by ultrasound)
* documented or suspected neuromuscular disease (thymoma, myasthenia, myopathies, muscular dystrophies, others)
* planned mechanical ventilation after surgery
* bilateral procedures
* lung separation with other method than DLT (e.g. difficult airway, tracheostomy)
* surgery in prone position
* persistent hemodynamic instability, intractable shock
* intracranial injury or tumor
* enrollment in other interventional study or refusal of informed consent
* pregnancy (excluded by anamnesis and/or laboratory analysis)
* esophagectomy, pleural surgery only, sympathectomy surgery only, chest wall surgery only, mediastinal surgery only, lung transplantation
* presence before induction of anaesthesia of one of the adverse events, listed as postoperative pulmonary complications (aspiration, moderate respiratory failure, infiltrates, pulmonary infection, atelectasis, cardiopulmonary edema, pleural effusion, pneumothorax, pulmonary embolism, purulent pleuritis, lung hemorrhage)
* documented preoperative hypercapnia > 45mmHg (6kPa)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2024-08 (Actual); Study Completion 2024-08 (Actual)

PRIMARY OUTCOMES:
The proportion of patients developing one or more postoperative pulmonary complications | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Mert Sentürk, Principal Investigator — Istanbul University Hospital
Locations (79):
- United States (3):
  - Tufts Medical Center, Boston, Massachusetts
  - NYC Cornell Medical College, New York, New York
  - Cleveland Clinic, USA, Cleveland, Ohio
- American Hospital Tirana, Tirana, Albania
- Medical University of Vienna, Vienna, Austria
- Brazil (3):
  - Hospital de Amor, Barretos, Barretos
  - Clinics Hospital from the Botucatu Medical School, University of Sao Paulo State, São Paulo
  - Sao Paulo Hospital, São Paulo
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- China (5):
  - First Affiliated Hospital of Guangzhou Medical University, China, Guangzhou
  - Anhui Provincial Hospital, First Aff. Hospital, University of Science and Technology of China, Hefei
  - Fudan University, Shanghai Cancer Center, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - West China Hospital Sichuan, Sichuan
- Croatia (2):
  - University Hospital Dubrava, Zagreb
  - University Hospital Zagreb, Zagreb
- Evangelistria Medical Center, Cyprus, Égkomi, Cyprus
- General University Hospital, Prague, Czechia
- Egypt (2):
  - Mansoura University Hospitals, Egypt, Al Mansurah
  - Tanta University Hospital, Tanta
- University Hospital of Dijon - François Mitterrand, Dijon, France
- Germany (7):
  - University Hospital Aachen, Aachen
  - Fachkrankenhaus Coswig, Coswig
  - Department of Anesthesiology and Intensive Care, Dresden University of Technology, Dresden
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Goettingen, Germany, Göttingen
  - University Hospital Magdeburg, Magdeburg
  - LMU Muenchen, München
- Greece (4):
  - Attikon University Hospital, Athens
  - Sotiria Chest Hospital, Athens
  - University Hospital of Heraklion, Heraklion
  - Patras University Hospital, Pátrai
- University of Debrecen, Department of anesthesiology and Intensive Care, Debrecen, Hungary
- Azadi Heart Center, Iraq, Duhok, Iraq
- Italy (8):
  - Arcispedale Sant'Anna, Ferrara
  - OORR Foggia, University of Foggia, Foggia
  - Ospedale Policlinico San Martino, Genova
  - AOU G.Martino, Messina
  - University Hospital Vanvitelli, Naples
  - University Hospital of Parma, Parma
  - University School of Medicine Campus Bio-Medico of Rome, Rome
  - University-Hospital of Udine, Udine
- Juntendo University Hospital, Tokyo, Japan
- Riga East University Hospital, Riga, Latvia, Riga, Latvia
- Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas, Mexico, Tlalpan, Mexico
- Netherlands (4):
  - Academic Medical Center Amsterdam, Amsterdam
  - VU medical center Amsterdam, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Radboud University Medical Centre Nijmegen, Nijmegen
- Institutul de Pneumoftiziologie Bucharest, Bucharest, Romania
- Department of Anesthesia, College of Medicine, King Saud University Medical City, Saudi-Arabia, Riyadh, Saudi Arabia
- Serbia (4):
  - Military Medical Academy, Belgrade
  - University Clinical centre of Serbia, Serbia, Belgrade
  - Clinical Center Nis, Clinic for anesthesia and intensive therapy, Niš
  - University of Novi Sad, Serbia, Novi Sad
- University Medical Centre Ljubljana, Ljubljana, Slovenia
- Spain (5):
  - Hospital Clínic. Universitat de Barcelona, Barcelona
  - Insular Hospital, Gran Canaria, Spain, Las Palmas de Gran Canaria
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario de La Ribera, Valencia
  - Hospital Álvaro Cunqueiro, Vigo
- University Hospital of Geneva, Geneva, Switzerland
- Taichung Veterans General Hospital, Taichung, Taiwan
- Turkey (Türkiye) (11):
  - Ankara Ataturk Chest Diseases And Chest Surgery Training and Research Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - University of Health Sciences, Bakırköy Dr. Sadi Konuk Training and Research Hospital, Turkey, Bakırköy
  - Acıbadem Mehmet Ali Aydınlar University, Istanbul
  - Istanbul Kartal Dr. Lutfi Kirdar Education and Research Hospital, Istanbul
  - Istanbul University, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - University of Health Science, Konya City Hospital, Turkey, Konya
  - Celal Bayar University Medical Faculty, Dept of Anesthesiology, Manisa
  - Mersin University Medical Faculty, Mersin
  - Pamukkale University Dinizli, Pamukkale
- United Kingdom (5):
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Golden Jubilee National Hospital, Clydebank
  - University Hospitals of Leicester, Leicester
  - St George's Hospital London, London
  - NIHS Sheffield Clinical Research Facility, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiss T, Wittenstein J, Becker C, Birr K, Cinnella G, Cohen E, El Tahan MR, Falcao LF, Gregoretti C, Granell M, Hachenberg T, Hollmann MW, Jankovic R, Karzai W, Krassler J, Loop T, Licker MJ, Marczin N, Mills GH, Murrell MT, Neskovic V, Nisnevitch-Savarese Z, Pelosi P, Rossaint R, Schultz MJ, Serpa Neto A, Severgnini P, Szegedi L, Vegh T, Voyagis G, Zhong J, Gama de Abreu M, Senturk M; PROTHOR investigators; Research Workgroup PROtective VEntilation Network (PROVEnet) of the European Society of Anaesthesiology (ESA). Protective ventilation with high versus low positive end-expiratory pressure during one-lung ventilation for thoracic surgery (PROTHOR): study protocol for a randomized controlled trial. Trials. 2019 Apr 11;20(1):213. doi: 10.1186/s13063-019-3208-8. PMID 30975217
- [Derived] Writing Committee; Steering Committee; PROTHOR Collaborative Group; PROtective VEntilation Network (PROVE Network) for the Clinical Trial Network of the European Society of Anaesthesiology and Intensive Care. Effects of intraoperative higher versus lower positive end-expiratory pressure during one-lung ventilation for thoracic surgery on postoperative pulmonary complications (PROTHOR): a multicentre, international, randomised, controlled, phase 3 trial. Lancet Respir Med. 2026 Jan;14(1):17-28. doi: 10.1016/S2213-2600(25)00330-3. Epub 2025 Nov 12. PMID 41240959
- See also: Trial Website — http://prothor.info
- Available data/document: Study Protocol — http://prothor.info

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT02963025/SAP_000.pdf